CLINICAL TRIAL: NCT00388271
Title: To Investigate if Alpha-blocker Therapy (Alfuzosin) Increases Stone Free Rates and Improves Pain Control After ESWL (Extra-corporeal Shock Wave Lithotripsy) for Renal and Ureteric Stones.
Brief Title: Use of Alfuzosin in Stone Treatment With ESWL
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Singapore General Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGH/URO/XTR001
Record Dates: First submitted 2006-10-13; First posted 2006-10-16 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Urinary Calculi
Keywords: Alpha-blocker; Alfuzosin; Xatral; ESWL
MeSH Terms: conditions — Urinary Calculi | interventions — alfuzosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): xatral
  Interventions: Drug: Alfuzosin (Xatral)
- 2 (Placebo Comparator): standard treatment
  Interventions: Drug: standard treatment

INTERVENTIONS:
Drug: Alfuzosin (Xatral) — standard treatment plus alfuzosin
  Arms: 1
Drug: standard treatment — standard treatment
  Arms: 2

SUMMARY:
Urinary tract stones may form in the kidneys or along the ureteric tracts and when left untreated, may result in complications such as pain, bleeding, infection and obstruction. ESWL (extra-corporeal shock wave lithotripsy) has been shown to be an effective and safe method of treatment for kidney and ureteric stones in-situ. In our centre, ESWL is done on an outpatient basis with oral pain killers in the weeks following treatment. Patients are also instructed to increase their fluid intake during this period to expedite the clearance of stone fragments. There have been studies to show that pain caused by stones is due to smooth muscle spasm along the ureters, possibly mediated by alpha-receptors. Alpha-blockers have been shown to improve the expulsion of stones and also improve pain relief when used alone, or together with ESWL treatment. In our study, we seek to investigate if alpha-blocker therapy (Alfuzosin) increases stone free rates and improves pain control after ESWL for renal and ureteric stones. The potential benefits include a higher rate of stone clearance and better pain control

DETAILED DESCRIPTION:
Urinary tract stones may form in the kidneys or along the ureteric tracts and when left untreated, may result in complications such as pain, bleeding, infection and obstruction. ESWL (extra-corporeal shock wave lithotripsy) has been shown to be an effective and safe method of treatment for kidney and ureteric stones in-situ. In our centre, ESWL is done on an outpatient basis with oral pain killers in the weeks following treatment. Patients are also instructed to increase their fluid intake during this period to expedite the clearance of stone fragments. Alpha1-adrenergic blockers have been shown to improve stone free rates in renal stones and lower ureteric stones. Tamsulosin has been the agent most commonly investigated. There have been no studies done to study the effectiveness of Alfuzosin in stone treatment. Alfuzosin has been shown to be effective in treating benign prostatic hypertrophy, and has a good safety profile. Deliveliotis et al has shown that alfuzosin improves symptoms and quality of life in patients with double-J stents.

This is a prospective, randomised, double-blind, placebo-controlled study involving patients undergoing ESWL for renal and ureteric stones. Exclusion criteria applies (please see below). The patients will be randomised into 2 groups: study VS control. Randomisation is done by using a computer generated list with block randomisation, assigning consecutive patients to either treatment arms. Our standard treatment is intravenous pethidine 50mg and intravenous maxolon 10mg at the onset of the ESWL session, followed by oral analgesics- NSAIDs with a gastroprotective agent. For this study, we will standardise all to oral naproxen 550mg BD with oral omeprazole 20mg BD. The study group will receive the standard treatment, with oral alfuzosin 10mg ON for 1 month, while the control group will receive a placebo. Patients will be given a diary in which to chart their pain scores, use of analgesics, episodes of pain, passage of stones, side-effects of the medications and complications of treatment. At the end of one month, all patients will be called back for review. Stone free status is ascertained with an X-ray, and the diary will be collected for further analysis.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients referred to our centre for ESWL treatment of renal or ureteric stones who give their informed consent.

Exclusion Criteria:

* Documented allergy or severe side effects to opioids/ NSAIDs/ Alfuzosin Severe hydronephrosis (on ultrasound or IVU) Radiolucent stones Urinary tract infections Previous pyeloureteral surgery Lower pole stones DJ stents in situ for stones Known renal/hepatic impairment or coagulopathy Pregnant Severe skeletal disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Reduction in pain score | 1 month
Reduction in use of analgesics | 1 month
stone free rate | 1 month

SECONDARY OUTCOMES:
Severe giddiness as a side-effect | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Tsung Wen Chong, MBBS, FRCS, Principal Investigator — SGH Urology
Locations (1):
- Urology Centre, Singapore, Singapore

REFERENCES:
- [Background] Gravina GL, Costa AM, Ronchi P, Galatioto GP, Angelucci A, Castellani D, Narcisi F, Vicentini C. Tamsulosin treatment increases clinical success rate of single extracorporeal shock wave lithotripsy of renal stones. Urology. 2005 Jul;66(1):24-8. doi: 10.1016/j.urology.2005.01.013. PMID 15992885